CLINICAL TRIAL: NCT06209450
Title: Sutured vs Suturless Mesh Fixation for Onlay Ventral Hernia Repair
Brief Title: Sutured vs Sutureless Mesh Fixation for Onlay Ventral Hernia Repair
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Khaled Mohammed Mahmoud Gadelhak, Assuit, Assiut University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Hernia
Record Dates: First submitted 2024-01-05; First posted 2024-01-17 (Actual); Last update posted 2024-01-17 (Actual); Status verified 2024-01

CONDITIONS: Ventral Hernia
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ventral hernia repair (Experimental)
  Interventions: Procedure: Ventral hernia repair with mesh fixation

INTERVENTIONS:
Procedure: Ventral hernia repair with mesh fixation — Sutured versus suturless mesh fixation

SUMMARY:
Comparison beta sutured and suturless mesh fixation for ventral hernia regarding recurrence rates and complications rate

DETAILED DESCRIPTION:
Ventral hernia repair is common procedure with over 250000 repairs each year in the unites states . Most ventral hernias are repaired using tension free type of repair using mesh that bridge the defect and reinforce the abdominal wall .

The mesh fixation technique has impact on recurrence rates,chronic pain and complications rates . Suturless ventral hernia repair with sealing agent fixation proved to be durable with comperable complication profile to other techniques.

ELIGIBILITY:
Inclusion Criteria:

* ventral hernia
* both sexes

Exclusion Criteria:

* obstructed or complicated ventral hernia
* incisional hernia
* recurrent hernia
* multiple ventral hernia
* large hernia more than 5 cm

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Estimated)
Dates: Start 2024-03-01 (Estimated); Primary Completion 2025-03-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Complications | One year after surgery
  Intraoperative and post operative complications occur due to technique used in study